CLINICAL TRIAL: NCT06634914
Title: 30-Day MoonBrew Sleep & Stress Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Efforia, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13210
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Sleep; Stress; Dietary Supplement

STUDY DESIGN:
Intervention Model Description: Single arm interventional.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Moonbrew 30 Days (Experimental): 30 Days of the Moonbrew Sleep cocktail consumed before bed.
  Interventions: Dietary Supplement: Moonbrew

INTERVENTIONS:
Dietary Supplement: Moonbrew — A blend of adaptogens with Chamomile, Rose, and Magnesium in a powdered form, designed to be mixed in liquid and consumed 2-3 hours before bed.

SUMMARY:
This study aims to assess how consuming MoonBrew each evening for 30 days impacts sleep quality and stress levels. Poor sleep and high stress often go hand-in-hand, worsening overall health. By using validated self-reported outcome measures, this study bridges the gap between anecdotal evidence and scientific proof (without requiring a connected health device), contributing valuable insights into natural solutions for better sleep.

DETAILED DESCRIPTION:
Poor sleep and high stress levels are pervasive issues affecting millions globally, leading to significant health problems. Research has consistently shown that poor sleep quality can exacerbate stress, while high stress levels can further disrupt sleep patterns. We have some great anecdotal evidence that suggests Moonbrew really works. This study aims to bridge the gap between anecdotal evidence and scientific evidence.

The aim of this study is to scientifically assess the impact of MoonBrew on sleep quality and stress levels using the PROMIS Sleep Disturbance Scale and NIH Toolbox® Item Bank v3.0 - Perceived Stress survey. Our objective is to determine whether regular consumption of MoonBrew can significantly improve sleep patterns and reduce stress over a 30-day period.

This study is significant as it seeks to provide scientific evidence on the efficacy of MoonBrew, a popular natural remedy, in enhancing sleep quality and reducing stress. Expected outcomes include improved sleep patterns and lower stress levels among participants. However, limitations include self-reported data and individual variations in response to MoonBrew. Nonetheless, the findings could pave the way for evidence-based recommendations and broader acceptance of natural sleep aids.

ELIGIBILITY:
Inclusion Criteria:

* US-based participants

Exclusion Criteria:

* allergies to mushrooms or adaptogens

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-10-14 (Estimated); Study Completion 2025-10-14 (Estimated)

PRIMARY OUTCOMES:
PROMIS Sleep Disturbance Scale | 30 days
  The PROMIS Sleep Disturbance Scale is a validated and widely used assessment tool developed as part of the Patient-Reported Outcomes Measurement Information System (PROMIS) initiative. It is designed to measure the severity of sleep disturbances and disruptions experienced by individuals. This scale includes a range of questions that assess the frequency and impact of various sleep-related issues, such as difficulty falling asleep, nighttime awakenings, and restless sleep. Healthcare professionals and researchers rely on this scale to better understand and quantify sleep problems in patients, enabling them to tailor interventions and treatment strategies to address sleep-related concerns effectively.
NIH Toolbox® Item Bank v3.0 - Perceived Stress (Ages 18+) - Fixed Form Survey: NIH Toolbox® Item Bank v3.0 - Perceived Stress (Ages 18+) - Fixed Form Survey Score | 30 Days
  The NIH Toolbox® Item Bank v3.0 - Perceived Stress (Ages 18+) - Fixed Form Survey is a standardized psychological assessment tool developed by the National Institutes of Health (NIH) to measure an individual's perceived stress levels. It is intended for use in adults aged 18 and above and is designed to provide a reliable and consistent measure of perceived stress. The fixed form survey includes a set of questions that assess an individual's subjective experiences related to stress, allowing healthcare professionals and researchers to gauge stress levels and its potential impact on overall health and well-being. This tool is a valuable resource for evaluating and monitoring stress in various clinical and research settings.

IPD SHARING:
Plan to Share IPD: Undecided